CLINICAL TRIAL: NCT03319680
Title: Prospective Randomized Multicenter Study to Demonstrate the Benefits of Hemodialysis Without Acetate (With Citrate): ABC-treat Study
Brief Title: Benefits of Hemodialysis With Citrate (ABC-treat) Study
Acronym: ABC-treat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Senefro (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABC-Treat
Record Dates: First submitted 2017-03-31; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Hemodialysis-Induced Symptom

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Citrate dialysate (Active Comparator): Hemodialysis with citrate dialysate during 16 weeks
  Interventions: Other: Citrate dialysate
- Acetate dialysate (No Intervention): Hemodialysis with acetate dialysate during 16 weeks

INTERVENTIONS:
Other: Citrate dialysate — Compare the effect of citrate dialysate with acetate dialysate
  Other Names: Acetate dialysate
  Arms: Citrate dialysate

SUMMARY:
Prospective randomized cross-over multicenter study to demonstrate the benefits of hemodialysis without acetate dialysate, with citrate.

32 weeks duration, in two phases. In the first, half of the patients started with citrate dialysate for 16 weeks and the other half with acetate dialysate, and then patients cross.

The primary objective is to analyze the effect of citrate dialysate on acid base balance decreasing chronic metabolic acidosis and avoiding / reducing post-dialytic alkalosis.

DETAILED DESCRIPTION:
Primary objective: to analyze the effect of citrate dialysate on acid base balance decreasing chronic metabolic acidosis and avoiding / reducing post-dialytic alkalosis.

Secondary objectives:

* Evaluate the effect of dialysate on the variation of calcium pre and post-dialytic, as well as on the parathormone (PTH)
* Assess the effect of dialysate on inflammation
* Assess the effect of dialysate on the Elimination of small and medium-sized molecules
* Assess the effect of dialysate on the tolerance to the hemodialysis sessions
* Assess the effect of dialysate on nutritional parameters

Patients: Adult patients dialysed three times per week for at least 3 months will be enrolled in 12 Spanish dialysis centres. Catheter as vascular access will be excluded.

Design: prospective randomized multicenter, cross-over trial of chronic haemodialysis patients to compare the effect of citrate dialysate with acetate dialysate.

Duration of study: 32 weeks, in two phases. Randomised to 16 weeks of hemodialysis with acetate followed by 16 weeks of citrate or 16 weeks of hemodialysis with citrate followed by 16 weeks of acetate. Each patient will serve as control of itself and there will be no changes in the pattern of dialysis during the study with the exception of the dialysate, following the usual pattern of work

ELIGIBILITY:
Inclusion Criteria:

* Outpatient conventional hemodialysis three times per week for at least three months.
* Arteriovenous fistula as vascular access
* Patients who have given their informed consent in writing.

Exclusion Criteria:

* Catheter as vascular access
* Allergy or intolerance to citrate
* Patients with sufficient cognitive impairment that would prevent the compression of information and informed consent.
* Inflammatory intercurrent diseases (chronic infections, autoimmune diseases or tumors) that can mask the results of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Effect of citrate dialysate on acid base status in hemodialysis patients measured by pH, BEecf and Bicarbonate at the end of HD session. | 32 weeks
  The anion gap will be calculated as: Anion gap = [Na+] - ([Cl-] + [CO3H-])

SECONDARY OUTCOMES:
Compare the effect of citrate dialysate with acetate dialysate on calcium level | 32 weeks
  Calcium (mg/dl) blood determination
Compare the effect of citrate dialysate with acetate dialysate on phosphate level | 32 weeks
  Phosphate (mg/dl) blood determination
Compare the effect of citrate dialysate with acetate dialysate on parathormone level. | 32 weeks
  Parathormone (pg/ml) blood determination
Inflammation status by blood determination of IL-6 | 32 weeks
  IL-6 (UI) blood determination
Inflammation status by blood determination of us-PCR | 32 weeks
  us-PCR (UI) blood determination
Inflammation status by blood determination of ERI | 32 weeks
  EPO Resistance Index (ERI) is calculated according to the following formula:
  ERI = EPO Dose (U/kg/week) / Hb (g/dl).
Effect of citrate dialysate on the hemodialysis elimination of small and medium-sized in molecules using reduction ratio (RR) of Urea | 32 weeks
  Urea reduction rates (RR) will be calculated as: RR (%) = [(Cpre - post)/Cpre] x 100.
  Where Cpre and Cpost are the concentrations of pre and post dialysis analyzed substances.
Effect of citrate dialysate on the hemodialysis elimination of small and medium-sized in molecules using reduction ratio (RR) of Beta2-microglobulin | 32 weeks
  β2m reduction rates (RR) will be calculated as: RR (%) = [(Cpre - post)/Cpre] x 100.
  Where Cpre and Cpost are the concentrations of pre and post dialysis analyzed substances.
  β2m concentrations at the end of the session will be corrected for concentration using a correction factor (FC) based on concentration of plasma proteins (PT): FC = PTpre/PTpost Where PTpre and PTpost are the concentrations of pre and post dialysis total proteins.
Effect of citrate dialysate on the tolerance to the hemodialysis sessions by determining number of intradyalitic hypotensions | 32 weeks
  Compare the effect of citrate dialysate with acetate dialysate on reduction ratio (RR) of hypotensive episodes (clinical syntoms) during the hemodialysis sessions
Effect of citrate dialysate on the nutritional parameters measured by biological parameters | 32 weeks
  Weight (Kg).
Effect of citrate dialysate on the nutritional parameters measured by biological parameters | 32 weeks
  Normalized-protein catabolism rate corrected by body weight (PCR-n) is calculated using the following formula: PCRn = PCR/weight (kg) PCR= (9.35×G) + (0.00028×V) G: generation of interdialytic urea: G = [(C3-C2)×V]/2646 is the generation of interdialytic urea C2 = urea concentration at the end of hemodialysis C3 = urea concentration at the start of the following hemodialysis session parameters

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Perez-Garcia, PhD, Principal Investigator — Nephrology department. Hospital universitario Infanta Leonor
Locations (12):
- Spain (12):
  - Hospital General de Castellón, Castellon, Castellón
  - Hospital del Henares, Coslada, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Universitario Santa Lucía, Cartagena, Murcia
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital de Galdakao, Usansolo, Vizcaya
  - Hospital Universitario de Guadalajara, Guadalajara
  - Universitary Hospital Infanta Leonor, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gabutti L, Lucchini B, Marone C, Alberio L, Burnier M. Citrate- vs. acetate-based dialysate in bicarbonate haemodialysis: consequences on haemodynamics, coagulation, acid-base status, and electrolytes. BMC Nephrol. 2009 Mar 5;10:7. doi: 10.1186/1471-2369-10-7. PMID 19265544
- [Background] Kossmann RJ, Gonzales A, Callan R, Ahmad S. Increased efficiency of hemodialysis with citrate dialysate: a prospective controlled study. Clin J Am Soc Nephrol. 2009 Sep;4(9):1459-64. doi: 10.2215/CJN.02590409. Epub 2009 Aug 6. PMID 19661218
- [Background] Bryland A, Wieslander A, Carlsson O, Hellmark T, Godaly G. Citrate treatment reduces endothelial death and inflammation under hyperglycaemic conditions. Diab Vasc Dis Res. 2012 Jan;9(1):42-51. doi: 10.1177/1479164111424297. Epub 2011 Nov 1. PMID 22045866
- [Background] Daimon S, Dan K, Kawano M. Comparison of acetate-free citrate hemodialysis and bicarbonate hemodialysis regarding the effect of intra-dialysis hypotension and post-dialysis malaise. Ther Apher Dial. 2011 Oct;15(5):460-5. doi: 10.1111/j.1744-9987.2011.00976.x. PMID 21974699
- [Background] Grundstrom G, Christensson A, Alquist M, Nilsson LG, Segelmark M. Replacement of acetate with citrate in dialysis fluid: a randomized clinical trial of short term safety and fluid biocompatibility. BMC Nephrol. 2013 Oct 9;14:216. doi: 10.1186/1471-2369-14-216. PMID 24103587
- [Background] Molina Nunez M, de Alarcon R, Roca S, Alvarez G, Ros MS, Jimeno C, Bucalo L, Villegas I, Garcia MA. Citrate versus acetate-based dialysate in on-line haemodiafiltration. A prospective cross-over study. Blood Purif. 2015;39(1-3):181-187. doi: 10.1159/000371569. PMID 25791278
- [Background] Kuragano T, Kida A, Furuta M, Yahiro M, Kitamura R, Otaki Y, Nonoguchi H, Matsumoto A, Nakanishi T. Effects of acetate-free citrate-containing dialysate on metabolic acidosis, anemia, and malnutrition in hemodialysis patients. Artif Organs. 2012 Mar;36(3):282-90. doi: 10.1111/j.1525-1594.2011.01349.x. Epub 2011 Sep 29. PMID 21954915
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593
- [Derived] de Sequera Ortiz P, Perez Garcia R, Molina Nunez M, Munoz Gonzalez RI, Alvarez Fernandez G, Merida Herrero E, Camba Caride MJ, Blazquez Collado LA, Alcaide Lara MP, Echarri Carrillo R; en representacion del grupo del estudio ABC-treat; Grupo del estudio ABC-treat. Prospective randomised multicentre study to demonstrate the benefits of haemodialysis without acetate (with citrate): ABC-treat Study. Acute effect of citrate. Nefrologia (Engl Ed). 2019 Jul-Aug;39(4):424-433. doi: 10.1016/j.nefro.2018.11.002. Epub 2019 Jan 24. English, Spanish. PMID 30686542
- See also: Sponsor web page — http://www.senefro.org/